CLINICAL TRIAL: NCT05645250
Title: Feasibility of a Newborn Screening for Spinal Muscular Atrophy (SMA) in France: DEPISMA Prefigurator Project in Grand Est and Nouvelle Aquitaine
Brief Title: Feasibility of a Newborn Screening for Spinal Muscular Atrophy (SMA) in France: DEPISMA Prefigurator Project in Grand-Est and Nouvelle-Aquitaine
Acronym: DEPISMA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8121
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-03

CONDITIONS: Feasibility of Neonatal Screening for Spinal Amyotrophy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Negatives cases
- Positive cases

SUMMARY:
Spinal muscular atrophy (SMA) is a genetic disease of the nervous system that affects about 1 in 7,0001.2 births and results in very high mortality for patients with the disease. There are about 120 new cases in France each year and an estimated total of 2500 patients. It is the leading cause of genetic mortality in children in France. Until 2017, no etiological treatment was available. Currently, three treatments have been approved and have authorizations in France. The current clinical developments in SMA show the importance of an early treatment for patients. 3. The identification of pre-symptomatic patients is therefore essential to improve the effectiveness of treatments on an individual level and to avoid any loss of chance, as well as to reduce the societal cost of disability for patients treated in post-symptomatic. Several countries in Europe and around the world have implemented regional pilot screening programs for the disease. The screening test is based on a molecular genetic analysis that has been performed for many years, and which is highly reliable; there is currently no biochemical marker that can be used.

The objective of our project is to demonstrate the feasibility of neonatal screening for spinal amyotrophy in two French regions before being able to propose to extend it to the whole of France. The management of all screened patients will be decided outside the pilot study, by the existing national multidisciplinary consultation meeting, according to the best available standards of care and will be based on the national network of neuromuscular disease reference centers The objective of the project is not the evaluation of the efficacy of treatments or neonatal screening: these objectives are being studied by existing or otherwise ongoing studies around the world.

This project has been set up to be in line with the existing structures in France that are responsible for neonatal screening (via the regional neonatal screening centers (CRDN) and the regional perinatal networks) and for the management of rare diseases (via the neuromuscular disease reference centers and their FILNEMUS network). This project is performed in collaboration with AFM Telethon, Directorate of Health Care Supply, Regional Health Agency (ARS), FILNEMUS network, Novartis Gene Therapies, Roche Pharma AG,Biogen.

Investigator wish, as far as possible, to bring this study closer to real life and to be able to generate as much information as possible that can be used directly to prefigure the potential generalization of this screening strategy to the entire national territory.

ELIGIBILITY:
Inclusion Criteria:

* - Newborns born in the Grand-Est or Nouvelle Aquitaine regions during the study period
* Parent(s) or legal guardian(s) who do not object to "conventional" newborn screening
* Parent(s) or legal guardian(s) who give consent for newborn screening for SMA
* Child with health coverage

Exclusion Criteria:

* Parent(s) under curators or guardianship

Ages: 1 Day to 5 Days | Sex: All
Age Groups: Child
Study Population: Participation in the study will be offered to the parents of all newborns meeting the inclusion criteria, along with the standard national newborn screening program
Sampling Method: Non-Probability Sample
Enrollment: 220000 (Estimated)
Dates: Start 2022-12-13 (Actual); Primary Completion 2024-12-12 (Estimated); Study Completion 2024-12-12 (Estimated)

PRIMARY OUTCOMES:
Completeness of screening for spinal muscular atrophy | 2 years
  The completeness of screening for spinal muscular atrophy will be measured by the ratio of the number of tests collected in our study to the number of births in the maternity units included in the study. This rate will also be complemented by the ratio of the number of tests collected in our study to the number of births recorded by the civil registry in the two study regions. These rates will be compared to the completeness rates observed in other European studies.
Time frames calculation | 2 years
  The time required from birth to management in a multidisciplinary consultation meeting according to the existing procedure (videoconference or electronic discussion group) (=TRCP) and the time from birth to the effective start of treatment = (TTTT) will be calculated from the data collected in the Case Report Form (CRF) for positive cases. These times will be compared with the times observed in comparable programs worldwide. The time to effective treatment initiation will be compared to the 6-week postnatal target used in the pre-symptomatic clinical trials.

SECONDARY OUTCOMES:
Evaluation of screening costs | 2 years
  The study will distinguish between costs related to screening and those related to the follow-up and evaluation of the pilot (cost related to the clinical research status). Within the costs related to screening, it will distinguish between fixed costs (which do not depend on the number of screenings) and variable costs (depending on the number of screenings).

CONTACTS AND LOCATIONS:
Overall Officials: Vincent LAUGEL, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (39):
- France (39):
  - Ch de Colmar - Hôpital Louis Pasteur, Colmar, Alsace
  - Hôpital Albert Schweitzer - Clinique Du Diaconat de Colmar, Colmar, Alsace
  - Ch de Haguenau, Haguenau, Alsace
  - Clinique Diaconat Fonderie de Mulhouse, Mulhouse, Alsace
  - Hôpital Emile Muller, Mulhouse, Alsace
  - Ch Ste Catherine, Saverne, Alsace
  - Cmco Chru de Strasbourg, Schiltigheim, Alsace
  - Ch de Selestat, Sélestat, Alsace
  - Clinique Rhena, Strasbourg, Alsace
  - Clinique Ste Anne, Strasbourg, Alsace
  - Chic de La Lauter, Wissembourg, Alsace
  - POLYCLINIQUE BEZANNES/Courlancy, Bezannes, Champagne Ardennes
  - CHIna HOPITAL MANCHESTER, Charleville-Mézières, Champagne Ardennes
  - Ch de Chaumont, Chaumont, Champagne Ardennes
  - Ch de Chalons En Champagne, Châlons-en-Champagne, Champagne Ardennes
  - Ch Epernay, Épernay, Champagne Ardennes
  - Chu Reims Höpital Maison Blanche, Reims, Champagne Ardennes
  - Groupement Hospitalier Aube Marne, Romilly-sur-Seine, Champagne Ardennes
  - Ch Genevieve Anthonioz de Gaulle, Saint-Dizier, Champagne Ardennes
  - Ch Troyes, Troyes, Champagne Ardennes
  - Ch Emile Durckheim, Épinal, Lorraine
  - Ch Marie Madeleine, Forbach, Lorraine
  - Ch de Luneville, Lunéville, Lorraine
  - Clinique Claude Bernard, Metz, Lorraine
  - Ch de Mont St Martin, Mont-Saint-Martin, Lorraine
  - Chru Nancy-Maternite, Nancy, Lorraine
  - Polyclinique Majorelle de Nancy, Nancy, Lorraine
  - Chic L'Ouest Vosgien Site Neufchateau, Neufchâteau, Lorraine
  - Ch de Remiremont, Remiremont, Lorraine
  - Clinique St Nabor, Saint-Avold, Lorraine
  - Ch St Charles, Saint-Dié, Lorraine
  - Ch de Verdun St Mihiel Hôpitalst Nicolas, Saint-Mihiel, Lorraine
  - Ch Saint Nicolas, Sarrebourg, Lorraine
  - Ch de Sarreguemines Hôpital Robert Pax, Sarreguemines, Lorraine
  - Chr Metz Thionville Hôpital de Mercy, Thionville, Lorraine
  - Hôpital Bel Air - Chr Metz -Thionville, Thionville, Lorraine
  - Ch St Charles, Toul, Lorraine
  - Ch de Briey- Hôpital Maillot, Briey
  - Vincent LAUGEL, Strasbourg

IPD SHARING:
Plan to Share IPD: No